CLINICAL TRIAL: NCT06205758
Title: Efficacy and Safety Prediction of Milrinone or Levosimendan as Initial Inotropic Drug Therapy in Patients With Acute and Advanced Heart Failure With Renal Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yi Han (Other)
Collaborators: Qianfoshan Hospital (Other)
Responsible Party: Sponsor-Investigator, Yi Han, Associate professor of pharmacy, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: LM001
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Levosimendan; Milrinone; Efficacy; Safety
Keywords: Acute and advanced heart failure; Milrinone; Levosimendan; renal insufficiency
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To evaluate the efficacy and safety of levosimendan and milrinone in the treatment of with acute heart failure with or without renal dysfunction;
2. Predictive modeling of the efficacy and safety of levosimendan and milrinone.

DETAILED DESCRIPTION:
By comparing the safety and efficacy of milrinone with levosimendan as an initial inotropic agent for the treatment of patients with acute heart failure with or without abnormal renal function, a preliminary efficacy and safety prediction model was developed for levosimendan and milrinone based on the basic characteristics of the patients and the level of renal function.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Patients who were clearly diagnosed with heart failure ( cardiac insufficiency ) and LVEF(Left Ventricular Ejection Fraction) < 50 %, and were judged by the physician to need and agree to use levosimendan or milrinone to maintain hemodynamic stability

Exclusion Criteria:

* chronic heart failure and New York Heart Association ( NYHA ) class I ~ II
* Complicated with infective endocarditis, aortic dissection, severe liver dysfunction ( child-pugh C ), severe renal insufficiency ( CrCl < 30 ml / min ), hypertrophic obstructive cardiomyopathy, ventricular assist device or surgical cardiac surgery within 30 days before the use of levosimendan
* Patients with severe ventricular arrhythmia 1 within 24 hours before levosimendan and systolic blood pressure 100 times / min within 2 hours before levosimendan
* During hospitalization, other positive inotropic drugs 2 were used when levosimendan was intravenously pumped or dripped, excluding the use of catecholamines for rescue
* received positive inotropic drug 2 treatment in the last 30 days
* Lack of serum creatinine, brain natriuretic peptide or brain natriuretic peptide precursor, serum total bilirubin, cardiac ultrasound baseline ( within 14 days before using levosimendan ) data
* pregnant and lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute heart failure (AHF), including new-onset acute heart failure AHF and acute decompensated chronic heart failure (ADHF), is usually associated with either mild or severe renal impairment. Deterioration of renal function can lead to a serious prognosis. Milrinone and levosimendan are the most commonly prescribed inotropic drugs with preclinical and clinical evidence of their renoprotective effects.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse outcome events | 30-days
  Adverse outcome events (within 30 days) included mortality, unplanned readmission, transfer to ICU, and resuscitation.

OTHER OUTCOMES:
Incidence of adverse reactions | 30-days
  Incidence of adverse reactions, including headache, hypotension, and cardiac arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Han, doctorate, Principal Investigator — First Affiliated Hospital of Shandon
Locations (1):
- First Affiliated Hospital of Shandong First Medical University ( Qianfoshan Hospital of Shandong Province ), Jinan, Shandong, China